CLINICAL TRIAL: NCT07012902
Title: The Interaction Between Remimazolam and Etomidate During Induction of General Anesthesia Was Studied by Isoradiometric Analysis
Brief Title: Relationship Between Remimazolam and Etomidate in Induction of General Anesthesia
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Second Hospital of Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Zheng Guo, professor, Second Hospital of Shanxi Medical University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: yuewei20250519
Record Dates: First submitted 2025-05-19; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Induction Anesthesia; Drug Interactions
Keywords: Isoradiation analysis; etomidate; remimazolam
MeSH Terms: interventions — Etomidate; remimazolam

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group A (remimazolam induction group) (Experimental): The ED50 of group A was calculated by sequential method
  Interventions: Drug: Etomidate
- Group B (etomidate induction group) (Experimental): The ED50 of group B was calculated by sequential method
  Interventions: Drug: Remimazolam
- group C (0.25ED50 remimazolam +0.75ED50 etomidate) (Experimental): The ED50 of etomidate in group C were calculated by sequential method.
  Interventions: Drug: Remimazolam-etomidate
- Group D (0.5ED50 remimazolam +0.5ED50 etomidate) (Experimental): The ED50 of etomidate in group Dwere calculated by sequential method.
  Interventions: Drug: Remimazolam-etomidate
- Group E (0.75ED50 remimazolam +0.25 etomidate) (Experimental): The ED50 of etomidate in group E were calculated by sequential method.
  Interventions: Drug: Remimazolam-etomidate

INTERVENTIONS:
Drug: Etomidate — Group A was induced with etomidate, the initial dose was 0.120mg/kg, and the ratio of adjacent doses was 1:0.6
  Arms: Group A (remimazolam induction group)
Drug: Remimazolam — Group B was induced with remimazolam, the initial dose was 0.20mg/kg, and the ratio of adjacent doses was 1:0.8
  Arms: Group B (etomidate induction group)
Drug: Remimazolam-etomidate — In group C, 0.25ED50 remimazolam +0.75ED50 etomidate was used as the initial measurement In group D, 0.5ED50 remimazolam +0.5ED50 etomidate was used as the initial measurement In group E, 0.75ED50 of remimazolam +0.25ED50 of etomidate was used as the initial measurement
  Arms: Group D (0.5ED50 remimazolam +0.5ED50 etomidate); Group E (0.75ED50 remimazolam +0.25 etomidate); group C (0.25ED50 remimazolam +0.75ED50 etomidate)

SUMMARY:
In modern anesthesia practice, anesthesiologists often need to choose a combination of multiple drugs according to the specific conditions and surgical needs of patients, which can not only achieve more fine anesthesia management, but also improve perioperative safety and patient comfort. In clinical practice, anesthesiologists will use etomidate combined with a small dose of remimazolam for anesthesia induction to obtain more stable hemodynamics, prevent intraoperative awareness, and relieve anxiety.However, what is the best dose ratio of etomidate combined with remimazolam, the current literature does not give clear indicators.

DETAILED DESCRIPTION:
The experiment was divided into two steps. Step 1: Patients were randomly divided into group A (remimazolam induction group) and group B (etomidate induction group) according to the random number table, and group A was selected according to the literature. In group B, the initial dose was 0.2mg/kg, and 0.120mg/kg, and the ratio of successive doses was 1:0.8 and 1: 0.6, the ED50 of group A and group B was calculated by the sequential method, and the calculated remimazolam and etomidate were used as the initial doses of subgroups Step 2: According to the random number table, the patients were divided into group C (0.25ED50 remimazolam +0.75ED50 etomidate), group D (0.5ED50 remimazolam +0.50ED50 etomidate), group E (0.75ED50 remimazolam +0.25ED50 etomidate), and the dose of remimazolam in each group was fixed. The ED50 of etomidate in group C, group D and group E were calculated by sequential method.

Anesthesia methods: One hundred and twenty-five patients of both sexes, aged 18-60 yr, of American Society of Anesthesiologists physical status I-II, BIM: 18-30kg/m2, undergoing general anesthesia in the Second Hospital of Shanxi Medical University, were selected. Before operation, the patients were required to fast and drink, and had not received special preoperative medication. After the patient entered the room, blood pressure, heart rate, oxygen saturation and BIS were monitored and oxygen inhalation was given to the mask for 5L/min. After the tripartite verification was correct, intravenous access was established in the patient's upper limb, fluid infusion was opened, anesthesia was induced, remimazolam and etomidate were injected directly and slowly intravenously, and remimazolam and etomidate were injected for more than 10s according to the dosage of each group. Two drugs were injected at an interval of 10s or more. After the completion of one drug injection, 5ml normal saline was used to flush the tube, and the score was scored 2 minutes after intravenous injection. BIS value of 45-60 was considered as a positive response, and the dose gradient of the next patient was reduced. The observation was calculated as the first patient with positive to negative turning point, and the observation ended when the next patient with positive to negative reaction at the seventh turning point. The secondary outcome measures were the incidence of adverse reactions, changes in heart rate and blood pressure. At the end of the observation, if the patient showed a negative reaction, 0.08mg/kg etomidate was added for sedation, and then sufentanil and rocuronium were given for tracheal intubation in turn, and then surgery was performed.The demographic data of the patients were collected, including: gender, age, height, weight, BIM Statistical methods: probit model was used to calculate ED50 of each group, and the drug correlation coefficient was introduced as 1/(actual dose of remimazolam/ED50 of remimazolam + actual dose of etomidate/ED50 of etomidate). The measurement data with normal distribution were expressed as mean ± standard deviation (x±s). The measurement data with normal distribution between group A and group B were compared by two independent sample t test, and the comparison between group C, group D and group E was compared by one-way analysis of variance. Graphpad prism software was used to make five groups of sequential experimental plots and iso-radiation analysis plots when P<0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Both sexes
2. aged 18-60 yr
3. ASA physical status I-II
4. BIM: 18-28kg/m²

Exclusion Criteria:

1. allergic to remimazolam and etomidate
2. in pregnancy or lactation
3. serious cardiovascular diseases, long-term alcoholism
4. used sedative drugs or opioids within 24 hours
5. severe mental illness and myasthenia gravis -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-06-12 (Estimated); Primary Completion 2025-06-19 (Estimated); Study Completion 2025-07-19 (Estimated)

PRIMARY OUTCOMES:
The ED50 value of etomidate in Group A | one week
  The sequential method was used to calculate the median effective dose of etomidate in group A. When the patient's BIS value was between 45 and 60, it was considered a positive response. For the next patient, the dose was reduced by one dose gradient; conversely, if it was a negative response, the dose was increased by one dose gradient. The observation was stopped when the first patient reached the positive-negative turning point, and the next patient with the positive-negative reaction was reached for the seventh turning point. The ED50 of each group was calculated using the probit model.
The ED50 value of Remimazolam in Group B | one week
  The sequential method was used to calculate the median effective dose of remimazolam in group B. A positive reaction was defined as a patient's BIS value ranging from 45 to 60. For the next patient, the dose was reduced by one dose gradient if it was a positive reaction, and increased by one dose gradient if it was a negative reaction. The observation was stopped when the next patient with the 7th positive-negative reaction point was reached. The ED50 of each group was calculated using the probit model.
Group C D E: etomidate ED50 | three weeks
  The sequential method was adopted to calculate the median effective dose of etomidate for groups C, D, and E separately. A patient was considered to have a positive response if their BIS value was between 45 and 60. For the next patient, the dose was reduced by one dose gradient if it was a positive response, and increased by one dose gradient if it was a negative response. The observation was ended when the next patient with the 7th positive-negative response was reached. The ED50 of each group was calculated using the probit model.
Isoradiation pattern | 24 hours
  The ED50 determined for groups A and B was plotted on the isoradiogram. The ED50 of etomidate and its 95% confidence interval were plotted on the horizontal axis, and the ED50 of remimazolam and its 95% confidence interval were plotted on the vertical axis. The two ED50 were connected to form an additive line, and the confidence interval was connected to form an additive line with 95% confidence interval. When the two drugs were used together, the effect intensity of the compound drugs fell on the additive line (or within the confidence interval), indicating that the two drugs had additive effect. On the left side of the addition line and confidence interval, it indicated that the two drugs had synergistic effect. If it falls on the right side, it is antagonistic.
drug correlation coefficient | 24 hours
  The drug correlation coefficient = 1/(actual dose of remimazolam/ED50 of remimazolam + actual dose of etomidate/ED50 of etomidate).

SECONDARY OUTCOMES:
muscle tremor | 5 weeks
  Side effects of etomidate
Bradycardia | 5 weeks
  The heart rate was less than 45 beats per minute
hypotension | 5 weeks
  Blood pressure is lower than the baseline by 20%.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Hospital of Shanxi Medical University, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: No